CLINICAL TRIAL: NCT02376205
Title: The Effectiveness of Postoperative Local Retropharyngeal Space Anesthetic to Reduce Dysphagia After Anterior Cervical Discectomy and Fusion Surgery
Brief Title: Anesthetic to Reduce Dysphagia After Anterior Cervical Discectomy and Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justin Parker Neurological Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: JPNI-4
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Dysphagia
Keywords: Anterior Cervical Discectomy and Fusion; Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Bupivacaine; Solutions; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine hydrochloride 0.5% solution (Experimental): Bupivacaine hydrochloride 0.5% 10 mL solution poured into the retropharyngeal space intraoperatively before wound closure during anterior cervical discectomy and fusion procedure
  Interventions: Drug: bupivacaine hydrochloride 0.5% solution
- 0.9% NaCl solution (Placebo Comparator): 0.9% NaCl 10 mL solution poured into the retropharyngeal space intraoperatively before wound closureduring anterior cervical discectomy and fusion procedure
  Interventions: Drug: 0.9% NaCl solution

INTERVENTIONS:
Drug: bupivacaine hydrochloride 0.5% solution — 10mL will be poured into the retropharyngeal space intraoperatively during anterior cervical discectomy and fusion procedure
  Other Names: Marcaine
  Arms: bupivacaine hydrochloride 0.5% solution
Drug: 0.9% NaCl solution — 10mL will be poured into the retropharyngeal space intraoperatively during anterior cervical discectomy and fusion procedure
  Other Names: Saline
  Arms: 0.9% NaCl solution

SUMMARY:
The main objective of this study is to analyze the effects of local anesthetic application into the retropharyngeal space and its ability to reduce dysphagia symptoms and/or occurrence rates in patients undergoing anterior cervical discectomy and fusion.

DETAILED DESCRIPTION:
The patients will be randomly assigned into one of the two groups to receive either bupivacaine hydrochloride 0.5% solution if they are randomized to the treatment group or 0.9% NaCl solution if they are randomized to the control group. These solutions will be poured into the retropharyngeal space intraoperatively before wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 y.o.
* Patients undergoing one- or two-level anterior cervical discectomy and fusion surgery for radiculopathy or myelopathy symptoms
* Patients are wiling and able to sign informed consent and complete questionnaires

Exclusion Criteria:

* More than 2-level ACDF surgeries
* Previous cervical spine surgery
* Surgeries for trauma, infection or tumor
* Known hypersensitivity reactions to bupivacaine hydrochloride or other amino-amide anesthetics (e.g. lidocaine)
* Known history of swallowing issues (e.g. dysphagia, odynophagia)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Reduction in dysphagia scores | 3 months
  Swallowing-Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Mason, MD, Principal Investigator — Boulder Neurosurgical Associates
Locations (1):
- Boulder Neurosurgical Associates, Boulder, Colorado, United States